CLINICAL TRIAL: NCT05654792
Title: Prognostic Factors in New-Onset Persistent Left Bundle Branch Block After Transcathether Aortic Valve Implantation
Brief Title: Prognostic Factors in NOP-LBBB After TAVI
Acronym: ProgNOP-LBBB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI163
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: transcatheter aortic valve implantation, aortic stenosis, permanent pacemaker, left bundle branch block, heart failure, cardiac dyssynchrony
MeSH Terms: conditions — Aortic Valve Stenosis; Bundle-Branch Block; Heart Failure | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NOP-LBBB: Patients with new-onset persistent left bundle branch block after transcatheter aortic valve implantation
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — Transcatheter aortic valve implantation in cases of severe aortic stenosis

SUMMARY:
The goal of this observational study is to find prognostic factors in patients with a new-onset persistent left bundle branch block (NOP-LBBB) after transcatheter aortic valve implantation (TAVI). The main question it aims to answer is:

Are there any factors influencing heart failure or death risk during the year following TAVI in patients with NOP-LBBB ? Participants will have data collection about TAVI procedure and clinical evolution during a one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* New-onset persistent left bundle branch block after transcatheter aortic valve implantation

Exclusion Criteria:

* Pre-existing left bundle branch block
* Pre-existing right bundle branch block
* Pre-existing permanent pacemaker
* Immediate procedural mortality (death ≤72 h post-procedure)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with transcatheter aortic valve implantation in University Hospital of Nancy between 2009 and 31/12/2021, and with left bundle branch block following transcatheter aortic valve implantation and persistent during hospitalisation
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalisation for heart failure or all-cause mortality | At one-year after transcatheter aortic valve implantation
  Hospitalisation for heart failure or all-cause mortality

SECONDARY OUTCOMES:
Hospitalisation for heart failure | At one-year after transcatheter aortic valve implantation
  Hospitalisation for heart failure
All-cause mortality | At one-year after transcatheter aortic valve implantation
  All-cause mortality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagaraja V, Raval J, Eslick GD, Ong AT. Transcatheter versus surgical aortic valve replacement: a systematic review and meta-analysis of randomised and non-randomised trials. Open Heart. 2014 Aug 12;1(1):e000013. doi: 10.1136/openhrt-2013-000013. eCollection 2014. PMID 25332780
- [Background] Hannan EL, Samadashvili Z, Stamato NJ, Lahey SJ, Wechsler A, Jordan D, Sundt TM 3rd, Gold JP, Ruiz CE, Ashraf MH, Smith CR. Utilization and 1-Year Mortality for Transcatheter Aortic Valve Replacement and Surgical Aortic Valve Replacement in New York Patients With Aortic Stenosis: 2011 to 2012. JACC Cardiovasc Interv. 2016 Mar 28;9(6):578-85. doi: 10.1016/j.jcin.2015.12.022. PMID 27013157
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Barbanti M, Gulino S, Costa G, Tamburino C. Pathophysiology, incidence and predictors of conduction disturbances during Transcatheter Aortic Valve Implantation. Expert Rev Med Devices. 2017 Feb;14(2):135-147. doi: 10.1080/17434440.2017.1282819. Epub 2017 Jan 21. PMID 28092726
- [Background] Urena M, Webb JG, Cheema A, Serra V, Toggweiler S, Barbanti M, Cheung A, Ye J, Dumont E, DeLarochelliere R, Doyle D, Al Lawati HA, Peterson M, Chisholm R, Igual A, Ribeiro HB, Nombela-Franco L, Philippon F, Garcia Del Blanco B, Rodes-Cabau J. Impact of new-onset persistent left bundle branch block on late clinical outcomes in patients undergoing transcatheter aortic valve implantation with a balloon-expandable valve. JACC Cardiovasc Interv. 2014 Feb;7(2):128-136. doi: 10.1016/j.jcin.2013.08.015. Epub 2014 Jan 15. PMID 24440024
- [Background] Houthuizen P, Van Garsse LA, Poels TT, de Jaegere P, van der Boon RM, Swinkels BM, Ten Berg JM, van der Kley F, Schalij MJ, Baan J Jr, Cocchieri R, Brueren GR, van Straten AH, den Heijer P, Bentala M, van Ommen V, Kluin J, Stella PR, Prins MH, Maessen JG, Prinzen FW. Left bundle-branch block induced by transcatheter aortic valve implantation increases risk of death. Circulation. 2012 Aug 7;126(6):720-8. doi: 10.1161/CIRCULATIONAHA.112.101055. Epub 2012 Jul 12. PMID 22791865
- [Background] Faroux L, Chen S, Muntane-Carol G, Regueiro A, Philippon F, Sondergaard L, Jorgensen TH, Lopez-Aguilera J, Kodali S, Leon M, Nazif T, Rodes-Cabau J. Clinical impact of conduction disturbances in transcatheter aortic valve replacement recipients: a systematic review and meta-analysis. Eur Heart J. 2020 Aug 1;41(29):2771-2781. doi: 10.1093/eurheartj/ehz924. PMID 31899484
- [Background] Regueiro A, Abdul-Jawad Altisent O, Del Trigo M, Campelo-Parada F, Puri R, Urena M, Philippon F, Rodes-Cabau J. Impact of New-Onset Left Bundle Branch Block and Periprocedural Permanent Pacemaker Implantation on Clinical Outcomes in Patients Undergoing Transcatheter Aortic Valve Replacement: A Systematic Review and Meta-Analysis. Circ Cardiovasc Interv. 2016 May;9(5):e003635. doi: 10.1161/CIRCINTERVENTIONS.115.003635. PMID 27169577
- [Background] Tsushima T, Main A, Al-Kindi SG, Dallan LAP, Wheat HL, Baeza CR, Pelletier MP, Arruda MS, Mackall JA, Thal SG, Ohno Y, Lee KH, Siqueira DA, Kaneko T, Harloff MT, Costa G, Barbanti M, Attizzani GF. Risk Stratification of New Persistent Left Bundle Branch Block After Transcatheter Aortic Valve Implantation. Am J Cardiol. 2022 Jul 15;175:80-87. doi: 10.1016/j.amjcard.2022.03.053. Epub 2022 May 18. PMID 35597627